CLINICAL TRIAL: NCT04085185
Title: A Phase 1a, Open-label, Dose-Escalation Study to Evaluate the Safety, Tolerability, and Initial Efficacy of IBI110 in Subjects With Advanced Malignant Tumors
Brief Title: A Study Evaluating the Safety, Tolerability, and Initial Efficacy of IBI110 in Subjects With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI110A101
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase Ia Dose-Escalation Stage:IBI110 (Experimental): Participants will be treated with escalating doses of IBI110 to determine the MTD.
  Interventions: Drug: IBI110
- Phase Ia Expansion Stage:IBI110 (Experimental): Participants will be enrolled in the expansion stage to better characterize the safety, tolerability, PK variability, and preliminary efficacy of IBI110 in different cancer types.
  Interventions: Drug: IBI110
- Phase Ib Dose-Escalation Stage:IBI110+ Sintilimab (Experimental): Participants will be treated with escalating doses of IBI110 in combination with a fixed dose of Sintilimab to determine the MTD.
  Interventions: Drug: IBI110+ Sintilimab
- Phase Ib Expansion Stage:IBI110+ Sintilimab (Experimental): Participants will be enrolled in the expansion stage to better characterize the safety, tolerability, PK variability, and preliminary efficacy of IBI110 in combination with Sintilimab in different cancer types.
  Interventions: Drug: IBI110+ Sintilimab

INTERVENTIONS:
Drug: IBI110 — Several dose levels will be evaluated for IBI110 administered as a single agent and in combination with Sintilimab. IBI110 will be given via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit. Those who discontinue treatment with single-agent IBI110 may receive combination treatment with IBI110 plus Sintilimab. Combination treatment may continue until disease progression or loss of clinical benefit.
  Arms: Phase Ia Dose-Escalation Stage:IBI110
Drug: IBI110 — IBI110 will be given with RP2D. IBI110 will be given via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit.
  Arms: Phase Ia Expansion Stage:IBI110
Drug: IBI110+ Sintilimab — IBI110: Several dose levels will be evaluated for IBI110 in combination with Sintilimab. IBI110 will be given via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit.
  Sintilimab: Sintilimab will be given as 200 mg via IV infusion on Day 1 of each 21-day cycle in combination with IBI110. Combination treatment may continue until disease progression or loss of clinical benefit.
  Arms: Phase Ib Dose-Escalation Stage:IBI110+ Sintilimab
Drug: IBI110+ Sintilimab — IBI110: IBI110 in combination with Sintilimab will be given with RP2D. IBI110 will be given via intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression or loss of clinical benefit.
  Sintilimab: Sintilimab will be given as 200 mg via IV infusion on Day 1 of each 21-day cycle in combination with IBI110. Combination treatment may continue until disease progression or loss of clinical benefit.
  Arms: Phase Ib Expansion Stage:IBI110+ Sintilimab

SUMMARY:
This is an open-label, dose escalation, Phase I study to evaluate the safety, tolerability, pharmacokinetics and efficacy of IBI110 in subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the ICF.
2. Adults 18 years of age or older.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy at least 12 weeks.
5. Adequate organ and bone marrow function.
6. Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumors and lymphomas that are refractory to standard therapy, or for which no standard therapy exists.
7. Measurable disease according to RECIST Version 1.1 in solid tumor.
8. Subjects (women of child-bearing potential and males) must be willing to use viable contraception method that is deemed effective by the investigator throughout the treatment period and for at least three months following the last dose of study drug. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:

1. Previous exposure to any anti-lag-3 antibody.
2. Participate in another interventional clinical study, except for the observational (non-interventional) clinical study or the survival follow-up phase of the interventional study.
3. Any investigational drugs received within 4 weeks prior to the first study treatment.
4. Receive the last dose of anti-tumor therapy within 4 weeks before the first dose of study therapy.
5. Immunosuppressive drugs were used within 4 weeks prior to the first administration of the study drug.
6. Medication requiring long-term systemic hormones or any other immunosuppression therapy.
7. Major surgical procedures (craniotomy, thoracotomy, or laparotomy) or unhealed wounds, ulcers, or fractures were performed within 4 weeks prior to the first dose of study therapy.
8. There were unrecovered toxicity (excluding hair loss or fatigue) according to NCI CTCAE v5.0 induced by previous antitumor therapy (24 weeks before the first dose of study), and there were unrecovered immune-related adverse events (irAE) associated with immunotherapy.
9. Previous immunotherapy, such as anti-PD-1 / anti-PD-L1 antibody or anti-CTLA4 antibody, was discontinued due to the presence of > grade 3 irAE.
10. Primary central nervous system (CNS) malignancy, or untreated/active CNS metastases, or leptomeningeal disease.
11. History of autoimmune disease , present active autoimmune disease or inflammatory diseases
12. Present or history of pulmonary diseases such as interstitial pneumonia, pneumoconiosis, drug-related pneumonia, pulmonary fibrosis, active pulmonary infection, severely impaired pulmonary function.
13. Positive human immunodeficiency virus (HIV) test.
14. Active hepatitis B or C, or tuberculosis.
15. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation. 16. History of gastrointestinal perforation and/or fistula at 6 months prior to study inclusion.

17.Hydrothorax, ascites, and pericardial effusion with clinical symptoms requiring drainage.

18.Known history of hypersensitivity to any components of the IBI110 or Sintilimab.

19.Uncontrolled complications of disease.

20.Other acute or chronic illness, mental illness, or abnormal laboratory test values that may increase the risk of study participation or administration of study drugs, or interfere with the interpretation of study results.

21.History of other primary malignancies. 22. Pregnant or nursing females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with AEs and SAEs | up to 2 years after enrollment
  To evaluate the safety and tolerability of IBI110 alone or in combination with Sintilimab [Adverse events (AEs), Serious Adverse Events (SAEs) ]
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | From Baseline to the end of Cycle 1
  To evaluate the safety and tolerability of IBI110 alone or in combination with Sintilimab.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | up to 2 years after enrollment
  The area under the curve (AUC) of serum concentration of the drug after the administration.
Pharmacokinetics: Cmax | up to 2 years after enrollment
  Maximum concentration (Cmax) of the drug after administration
Immunogenicity: Percentage of ADA positive subjects | up to 2 years after enrollment
  Immunogenicity: Number of Anti-Drug Antibodies (ADA) positive subjects will be counted and percentage of ADA positive subjects will be calculated to evaluate immunogenicity of IBI110.
Preliminary anti-tumor activity of IBI110 (Objective Response Rate) | up to 2 years after enrollment
  Objective Response Rate (ORR) is the percentage of Complete Response (CR) plus partial response (PR) assessed by RECIST v1.1 criteria for solid tumors and Lugano2014 criteria for lymphoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China

REFERENCES:
- [Derived] Wang Q, Xiong A, Mao C, Wang W, Cui J, Fang J, Zhuang W, Yang K, Zuo W, Yang J, Ye L, Zhang Z, Sheng Z, Liu Z, Wang D, Du X, Yi T, Long S, Xu N, Zhou C. Efficacy and safety of anti-LAG-3 IBI110 in combination with sintilimab and chemotherapy for advanced squamous non-small cell lung cancer: a randomized phase II study. Cancer Immunol Immunother. 2026 Jan 27;75(2):56. doi: 10.1007/s00262-026-04299-x. PMID 41591537
- [Derived] Mao C, Xiong A, Qian J, Wang W, Liu Y, Zhang T, Wu Z, Ni H, Lu J, Long S, Zhao L, Chen Y, Zhou C, Xu N. Dual inhibition of LAG-3 and PD-1 with IBI110 and sintilimab in advanced solid tumors: the first-in-human phase Ia/Ib study. J Hematol Oncol. 2024 Dec 31;17(1):132. doi: 10.1186/s13045-024-01651-5. PMID 39736787